CLINICAL TRIAL: NCT05124028
Title: A Study of Orelabrutinib in Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: A Study of Orelabrutinib in Patients With ITP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Clinical Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZXH-ITP2021
Record Dates: First submitted 2021-11-06; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Immune Thrombocytopenia
Keywords: Bruton's Tyrosine Kinase
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib (Experimental): Orelabrutinib 50mg po qd 6 weeks
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — 50mg po qd 6 weeks

SUMMARY:
This project was undertaken to evaluate the efficacy and safety of BTK inhibitor Orelabrutinib for the secondary treatment of adults with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a prospective trial of 10 adults with ITP in China. Orelabrutinib is administered as 50 mg po. qd for 6 weeks. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary refractory ITP
* Platelet counts <30×10^9/L or with bleeding symptoms
* Willing and able to sign written informed consent

Exclusion Criteria:

* Secondary thrombocytopenia
* Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit
* HIV infection or hepatitis B virus or hepatitis C virus infections
* Malignancy
* Severe medical condition (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
* Nursing or pregnant patients
* Patients who are deemed unsuitable for the study by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall response (OR) | 6 weeks
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-week follow-up.

SECONDARY OUTCOMES:
Complete response (CR) | 6 weeks
  Complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding.
Time to response | 6 weeks
  The time from starting treatment to time of achievement of Response.
Bleeding events | 6 weeks
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Side effects | 6 weeks
  Potential side effects include leukopenia, nausea and diarrhea, infectious diseases, etc .

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University Institute of Hematology
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No